CLINICAL TRIAL: NCT05929118
Title: The Impact of Aquatic Rehabilitation on Gait and Muscle Function in Patients After Anterior Cruciate Ligament Reconstruction.
Brief Title: The Effect of Aquatic Rehabilitation on Knee Function in Anterior Cruciate Ligament Reconstruction Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022158H
Record Dates: First submitted 2023-05-11; First posted 2023-07-03 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-01

CONDITIONS: Anterior Cruciate Ligament Reconstruction; Hydrotherapy; Gait; Muscle Function

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aquatic Rehabilitation (Experimental): Each group performed 70-90 minutes per session for a total of 6 interventions, all of which included warm-up activities, mobility training, strength training, functional exercise, and finishing activities. Each training was conducted 1-2 days apart, 2-3 times per week, and the training was completed within 2-3 weeks.
  Interventions: Other: Aquatic Rehabilitation
- Land-based Rehabilitation (Experimental): Each group performed 70-90 minutes per session for a total of 6 interventions, all of which included warm-up activities, mobility training, strength training, functional exercise, and finishing activities. Each training was conducted 1-2 days apart, 2-3 times per week, and the training was completed within 2-3 weeks.
  Interventions: Other: Land-based Rehabilitation

INTERVENTIONS:
Other: Aquatic Rehabilitation — Reviewing the existing literature studies and related books, and combining the post-operative rehabilitation process of ACLR with the opinions of experts from the China Aquatic Rehabilitation Association, the Aquatic rehabilitation program of this study was designed.
  Arms: Aquatic Rehabilitation
Other: Land-based Rehabilitation — Peking University Third Hospital Anterior Cruciate Ligament (ACL) Postoperative Rehabilitation Guidelines.
  Arms: Land-based Rehabilitation

SUMMARY:
The goal of this clinical trial is to compare the applicability and effectiveness of an aquatic rehabilitation training program with a conventional land-based rehabilitation program in terms of lower extremity biomechanics and knee function in Anterior Cruciate Ligament Reconstruction (ACLR) patients. The main questions it aims to answer are:

* Does aquatic rehabilitation accelerate the recovery of gait symmetry and muscle function in patients after ACLR？
* Previous studies have not uncovered the training characteristics of aquatic rehabilitation, which allow for training movements that cannot be performed on land, and it is unknown whether these different training movement characteristics are more effective for patients with ACLR.

Participants were randomly divided into an aquatic rehabilitation group (AR) and a land-based rehabilitation group (LR), and each group performed 70-90 minutes of training per session for a total of 6 sessions. This included warm-up activities, mobility training, strength training, functional exercises, and finishing activities. Each training session was conducted 1-2 days apart, 2-3 sessions per week, and the training was completed within 2-3 weeks.

DETAILED DESCRIPTION:
The experimental procedures of this study included collecting basic information about the subjects (age, height, weight, injury history, and surgery) and assessing muscle properties, degree of knee swelling, thigh circumference, knee flexion mobility, balance ability, gait, and the IKDC2000 score. Post-intervention testing was performed with the same testing procedures as the pre-intervention testing. The IKDC score was assessed again for one year after the intervention.

The results of all outcomes measured before and after the intervention were analyzed and calculated using IBM SPSS Statistics 26.0. The data were tested for normality using the Shapiro-Wilk test. For data conforming to a normal distribution, results are expressed as mean (Mean) and standard deviation (SD). An independent-samples t-test was used to compare whether there was a statistically significant difference in baseline and post-intervention values between the two intervention groups, and a paired-samples t-test was used to test whether there was a statistically significant difference before and after the intervention within each group. For data that did not conform to a normal distribution, results are expressed as median and interquartile range (IQR). The Mann-Whitney U test was used to compare baseline and post-intervention values between the two intervention groups, and the Wilcoxon signed-rank test was used to examine whether there was a statistically significant difference before and after the intervention within each group. Statistical significance was set at P < 0.05, and P < 0.01 was considered highly significant.

ELIGIBILITY:
Inclusion Criteria:

* Patients 4-8 weeks after unilateral ACL reconstruction surgery, or combined meniscus removal or resection, or 6-10 weeks after combined meniscus suturing after unilateral ACL reconstruction;
* No other lower extremity injury in the last 3 months, except for meniscal injury.

Exclusion Criteria:

* Contraindications related to underwater conditions such as open wounds, infectious diseases, history of neurological diseases (stroke, degenerative diseases of the central or peripheral nervous system, etc.), and being on psychotropic or anti-hypertensive drugs;
* Fear of water and inability to comply with experimental arrangements;
* History of ACL reconstruction surgery on the contralateral lower extremity and not more than half a year ago.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Stride Length Change | Each subject was tested before the first intervention training and after the sixth intervention training (on average 2-3 weeks after the first intervention).
  Kinovea 0.8.15 software was used for gait video calibration to analyze and calculate the stride length, which is the longitudinal linear distance between two consecutive heel touches on the same side of the foot during walking. The time, place, and testers of the test were kept consistent.
Step Length Change | Each subject was tested before the first intervention training and after the sixth intervention training (on average 2-3 weeks after the first intervention).
  Kinovea 0.8.15 software was used to calibrate the gait video to analyze and calculate the step length, which is the longitudinal linear distance between two points when the left and right heels touch the ground during walking. The time, place, and testers of the test were kept consistent.
Stride Length Time Change | Each subject was tested before the first intervention training and after the sixth intervention training (on average 2-3 weeks after the first intervention).
  Kinovea 0.8.15 software was used to calibrate the gait video to analyze and calculate the stride length, which is the time between two consecutive landings on the same side of the heel during walking. The time, place, and testers of the test were kept consistent.
Step Length Time Change | Each subject was tested before the first intervention training and after the sixth intervention training (on average 2-3 weeks after the first intervention).
  Kinovea 0.8.15 software was used to calibrate the gait video to analyze and calculate the step length time, which is the time between the two points where the left and right heels touch the ground during walking. The time, place, and testers of the test were kept consistent.
Single Support Phase Change | Each subject was tested before the first intervention training and after the sixth intervention training (on average 2-3 weeks after the first intervention).
  Kinovea 0.8.15 software was used to calibrate the gait video to analyze and calculate the single support phase, which is the time between the toe of one foot leaving the ground and the foot following the ground on that side during walking. The time, place, and testers of the test were kept consistent.
Oscillation Frequency Change | Each subject was tested before the first intervention training and after the sixth intervention training (on average 2-3 weeks after the first intervention).
  Oscillation Frequency (Hz) is the intrinsic pressure of the muscle, that is, the pressure carried by the muscle itself in the relaxed state or in the absence of voluntary contraction, and represents the muscle tone. The time, place, and testers of the test were kept consistent.
Mechanical Stress Relaxation Time Change | Each subject was tested before the first intervention training and after the sixth intervention training (on average 2-3 weeks after the first intervention).
  Mechanical Stress Relaxation Time (MSRT) is the time required for the muscle to return from its deformed state to its original state after active contraction or withdrawal of external pressure. The time, place, and testers of the test were kept consistent.
Creep Change | Each subject was tested before the first intervention training and after the sixth intervention training (on average 2-3 weeks after the first intervention).
  Creep (Deborah number) is the ratio of the mechanical stress release time to the time required for the muscle to reach maximum deformation by external force, SRT and Creep represent muscle viscosity. The time, place, and testers of the test were kept consistent.
Range of Motion Change | Each subject was tested before the first intervention training and after the sixth intervention training (on average 2-3 weeks after the first intervention).
  Active and passive Range of Motion in knee flexion. The time, place, and testers of the test were kept consistent.
2000 IKDC Subjective Knee Evaluation Form Change | Each subject was tested before the first intervention training and after the sixth intervention training (on average 2-3 weeks after the first intervention). Follow-up was performed again one year after the end of the intervention using the IKDC score.
  2000 IKDC Subjective Knee Evaluation Form is divided into three modules: knee symptoms (7 questions), motor activity (10 questions) and self-functional score (2 questions), where knee symptoms include frequency and degree of pain, stiffness, swelling, locking and instability; motor activity includes activity level, going up and down stairs, squatting, kneeling straight down, sitting and standing up with bent knees, running, jumping and landing on the affected limb, and quick starts and stops; and self-functional score includes pre-injury and current self-functional scores, graded from unable to perform daily activities (0 points) to unrestricted daily activities (10 points). The time, place, and testers of the test were kept consistent.
Stiffness Change | Each subject was tested before the first intervention training and after the sixth intervention training (on average 2-3 weeks after the first intervention).
  Stiffness indicates the resistance of a muscle to contraction or to an external force that deforms its initial shape. The time, place, and testers of the test were kept consistent.
Decrement Value Change | Each subject was tested before the first intervention training and after the sixth intervention training (on average 2-3 weeks after the first intervention).
  The Decrement (Dec) value represents a muscle's ability to return to its initial shape after the reduction or removal of an external force, with muscle elasticity being inversely proportional to the Dec value. A lower Dec value indicates greater muscle elasticity. The time, place, and testers of the test were kept consistent.

SECONDARY OUTCOMES:
Degree of Knee Swelling Change | Each subject was tested before the first intervention training and after the sixth intervention training (on average 2-3 weeks after the first intervention).
  The circumference of the knee joint was measured with a soft tape to indicate the degree of swelling of the knee joint. The subject was placed in a supine position with the lower extremities in a slightly flexed and relaxed position, and the hands were placed naturally on the side of the body. The medial and lateral femoral condyles were used as the midline of the knee joint, and the circumference of the knee joint enclosed by this midline was measured and recorded with the upper edge of the soft dipstick to reflect the swelling of the knee joint. The swelling effect of the intervention was reflected by the change in the circumference of the knee before and after training, and the difference in circumference between the two sides could reflect the degree of swelling. The time, place, and testers of the test were kept consistent.
Thigh Muscle Atrophy Change | Each subject was tested before the first intervention training and after the sixth intervention training (on average 2-3 weeks after the first intervention).
  Thigh circumference can indirectly indicate the strength of the knee flexor and extensor muscles by indirectly reflecting the cross-sectional area of the thigh muscles, so the circumference of the thigh at 10 cm above the patella was measured with a soft dermatome to reflect the muscle strength of the thigh, and the resulting atrophy index was calculated to reflect the degree of atrophy of the thigh. The time, place, and testers of the test were kept consistent.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Song, Doctor, Principal Investigator — Beijing Sport University
Locations (1):
- Beijing Sport University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No